CLINICAL TRIAL: NCT04078464
Title: Affective and Cognitive Responses to Acute Bouts of Aerobic Exercise, Mindfulness Meditation, and Combined Exercise and Meditation
Brief Title: Affective and Cognitive Responses to Acute Bouts of Physical Activity and Mindfulness Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Siobhan M Phillips, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00210138
Record Dates: First submitted 2019-08-20; First posted 2019-09-06 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Behavior
Keywords: Mindfulness; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: The order the participants participate in the 3 experimental conditions will be randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute Physical Activity + Mindfulness training (Experimental): 20 minutes of walking on a treadmill at a moderate pace while listening to a pre-recorded guided mindfulness meditation.
  Interventions: Other: Acute Physical Activity and Mindfulness Training Together
- Mindfulness training (Experimental): Participants will lie down and listen to a pre-recorded guided mindfulness meditation for 20 minutes.
  Interventions: Other: Mindfulness Training Alone
- Acute Physical Activity (Experimental): 20 minutes of walking on a treadmill at a moderate pace.
  Interventions: Other: Acute Physical Activity Alone

INTERVENTIONS:
Other: Mindfulness Training Alone — Participants will lie down and listen to a pre-recorded guided mindfulness meditation for 36 minutes.
  Arms: Mindfulness training
Other: Acute Physical Activity Alone — Physical activity will include a 6 minute stretching session, 1 minute transition to treadmill, 3 minute warm up at a participant chosen pace on the treadmill, 20 minutes of walking at a moderate pace at target heart rate, 3 minute cool down at 2.0-2.5 mph, 1 minute transition off treadmill and 2 minutes of stretching.
  Arms: Acute Physical Activity
Other: Acute Physical Activity and Mindfulness Training Together — Participants will listen to a pre-recorded mindfulness meditation which will guide them through a 6 minute stretching session, 1 minute transition to treadmill, 3 minute warm up at a participant chosen pace on the treadmill, 20 minutes of walking at a moderate pace at target heart rate, 3 minute cool down at 2.0-2.5 mph, 1 minute transition off treadmill and 2 minutes of stretching.
  Arms: Acute Physical Activity + Mindfulness training

SUMMARY:
The purpose of the present study is to investigate the benefits of mindfulness training during an acute bout of physical activity. We will compare the combination of mindfulness training and physical activity to mindfulness training alone and physical activity alone in three 20 minute sessions.

DETAILED DESCRIPTION:
We will investigate whether mindfulness training during a single bout (20 minutes) of physical activity influences ratings of perceived exertion, feeling states and physiological response (blood pressure and heart rate) during physical activity. Changes in affect and cognitive function pre- and post- physical activity bout will also be assessed. The effects of mindfulness training during an acute bout of physical activity will be compared to mindfulness training alone and acute physical activity alone. This research will contribute to larger questions of how to increase rates of physical activity in the general population and make physical activity more enjoyable.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in spoken and written English
* Have access to internet to complete baseline and post-study assessments

Exclusion Criteria:

* Respiratory, joint, or cardiovascular problems precluding physical activity participation
* Fail the Physical Activity Readiness Questionnaire (PAR-Q) and are unable to obtain physician consent to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Response of heart rate (beats per minute) to mindfulness training. | 36 minutes
  Heart rate will be measured using a polar heart rate monitor.and will be recorded every minute during the intervention.
Response of blood pressure (mm/Hg) to mindfulness training. | 36 minutes
  Blood pressure will be measured manually every 4 minutes during the intervention
Influence of mindfulness training on perceived exertion as measured by the Borg's Rating of Perceived Exertion scale (RPE). | 36 minutes
  Perceived exertion will be measured using Borg's Rating of Perceived Exertion scale. Participants will be asked how hard they perceive they are working every minute during the intervention on a scale from 6 to 20, with 6 being no work and 20 being working very, very hard.
Influence of mindfulness training feeling state as measured by the Feeling Scale (FS). | 36 minutes
  Participants will be asked to rate how they feel, using the Feeling Scale (FS), every minute during the intervention. The scale ranges from -5 to +5 with -5 being very bad and +5 being very good.

SECONDARY OUTCOMES:
Intervention effect on mindfulness as measured by the State Mindfulness Scale | 36 minutes
  Mindfulness will be assessed using the State Mindfulness Scale, after the intervention, at each study visit. Participants will rate their awareness of physical sensations and mental events (emotions, thoughts) on a scale of 1-5. 1=not at all, 2= a little, 3=somewhat, 4=well, 5=very well. There are 21 items on the scale. A higher score is indicative of greater mindfulness.
Intervention effect on affect as measured by the Positive and Negative Affect Schedule (PANAS). | 36 minutes
  Affect will be measured using the Positive and Negative Affect Schedule (PANAS) before and after the intervention. Participants rate how they have felt this week, in response to words describing feelings, on a scale from 1-5; 1=Very Slightly or Not at all, 2= A Little, 3= Moderately, 4= Quite a bit, 5= Extremely. PANAS is divided into two sub-scales for positive and negative affect. Positive affect scores range from 10-50 with a higher score representing higher levels of positive affect. Negative affect scores also range from 10-50 with lower scores representing lower levels of negative affect.
Intervention effect on anxiety will be assessed using the State Trait Anxiety Inventory (STAI) | 36 minutes
  Anxiety will be measured using the State Trait Anxiety Inventory (STAI) before and after the intervention. Participants will rate how they feel right now, in response to 20 statements about how people may feel, on a scale of 1-4; 1=Not at all, 2= Somewhat, 3=Moderately So, 4= Very much so. Total score ranges between 20 and 80 with 20-37 being no or low anxiety, moderate anxiety=38-44, and high anxiety=45-80.
Intervention effect on cognition as measured by NIH Toolbox Flanker Inhibitory Control and Attention Test (Flanker) | 36 minutes
  Participants will complete the NIH toolbox Flanker Inhibitory Control and Attention Test on an iPad before and after the intervention. The Flanker test is scored as a combination of the accuracy score and reaction time score. Score range is 0-10 with a higher score indicating a better performance.
Intervention effect on cognition as measured by NIH Toolbox List Sorting Working Memory Test. | 36 minutes
  Participants will complete the NIH Toolbox List Sorting Working Memory Test on an iPad before and after the intervention. The test is scored as the total number of items correctly recalled and sequenced. Score range is 0-26, with a higher score indicating a better performance.
Intervention effect on cognition as measured by NIH Toolbox Dimensional Change Card Sort Test. | 36 minutes
  Participants will complete the NIH Toolbox Dimensional Change Card Sort Test on an iPad before and after the intervention. The test is a measure of cognitive flexibility. The test is scored as a combination of the accuracy score and reaction time score. Score range is 0-10 with a higher score indicating a better performance.
Intervention effect on cognition as measured by NIH Toolbox Pattern Comparison Processing Speed Test | 36 minutes
  Participants will complete the NIH Toolbox Pattern Comparison Processing Speed Test on an iPad before and after the intervention. The test is scored as the sum of the number of items answered correctly in 90 seconds. Score range is 0-130. Higher scores indicate faster speed of processing.
Intervention effect on cognition as measured by NIH Toolbox Picture Sequence Memory Test. | 36 minutes
  Participants will complete the NIH Toolbox Picture Sequence Memory Test before and after the intervention. The Picture Sequence Memory Test measures episodic memory; cognitive processes involved in the acquisition, storage, and retrieval of new information. Participants are given credit for each adjacent pair of pictures they correctly place, up to 17 points. A higher score indicates a better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States